CLINICAL TRIAL: NCT04152213
Title: The Effects of Low Glycemic Index (GI) Diet on Cardiometabolic Outcomes Among Obese Chinese Adults: A Randomized Controlled Trial
Brief Title: The Effects of Low Glycemic Index (GI) Diet on Cardiometabolic Outcomes Among Obese Chinese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Leung Lai Yin, Doctoral Student, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00000000
Record Dates: First submitted 2019-10-30; First posted 2019-11-05 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Central Obesity
Keywords: Chinese adult; obesity; low glycemic index diet; cardiometabolic
MeSH Terms: conditions — Obesity; Obesity, Abdominal

STUDY DESIGN:
Intervention Model Description: prospective, two-arm randomized-controlled trial
Who Masked: Outcomes Assessor
Masking Description: Research assistants who have no knowledge about group allocation and study's objectives, will collected the post-intervention data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low GI diet group (Experimental): The components of the Low GI diet group include:
  (1) A one-off, 60-minute, face-to-face, educational session conducted by the research nurse for GI knowledge input. (2) An informational booklet will be given out during the education session. (3) Three follow-up telephone calls of fifteen minutes will be conducted by the research nurse at the 2nd, 5th , and 8th weeks after completing the face-to-face education session.
  Interventions: Behavioral: Low GI diet
- Control group (Placebo Comparator): The components of the control group include:
  (1) Pamphlets from the Department of Health about obesity and a balanced diet based on the food pyramid will be distributed. (2)Three follow-up telephone calls of fifteen minutes will be conducted by the research nurse at the 2nd, 5th , and 8th weeks after receiving the pamphlets.
  Interventions: Behavioral: Low GI diet

INTERVENTIONS:
Behavioral: Low GI diet — This educational session will cover information on obesity, complications of obesity, the benefit of weight loss, the glycemic index and its associated low GI diet, a food-exchange table including high- to low-GI foods, and self-decision in food choices. The dietary advice will be based on the standard food pyramid for the conventional Chinese diet as promoted by the Hong Kong Department of Health, with an emphasis on the selection of low-GI products. Practical tips will be given such as the selection of low-GI rice and rice products, the impact of cooking methods (including cooking time, cooking conditions, and cooking liquid volume) on rice GI, intervention to reduce the GI of rice, and listing low-GI food options and meal plans.

SUMMARY:
The aim of this study is to investigate the effects and the acceptability of low GI diet versus a conventional healthy diet on the BMI and other cardiometabolic risk factors of obese Chinese adults in Hong Kong.

DETAILED DESCRIPTION:
29.9% of persons aged 15-84 in Hong Kong are obese. Obesity poses significant detrimental consequences for one's health. Obese patients have an increased risk of mortality when compared with people with normal BMI. Obesity results in arterial hypertension, hyperlipidaemia, heart disease and type 2 diabetes. Low GI diets have been investigated for their impact on weight control. Evidence showed that low GI diets were effective in lowering body mass index. However, the evidence was usually generated from Western populations, thus excluding the influence of Chinese culture on diet.The aim of this study is to investigate the effects and the acceptability of low GI diet versus a conventional healthy diet on the BMI and other cardiometabolic risk factors of obese Chinese adults in Hong Kong.

A prospective, two-arm randomized-controlled trial will be conducted to examine the effect of a low GI diet education program on cardiometabolic outcomes in Chinese adults with obesity. The intervention group will receive a low GI diet education, including a one-off, 60-minute, face-to-face, educational session conducted by the research nurse for GI knowledge input. An informational booklet will be given out during the education session.Three follow-up telephone calls of fifteen minutes will be conducted by the research nurse at the 2nd, 5th , and 8th weeks after completing the face-to-face education session. While the control group will receive an education pamphlets on obesity and balanced diet.Three follow-up telephone calls of fifteen minutes will be conducted by the research nurse at the 2nd, 5th , and 8th weeks after receiving the pamphlets.

At baseline, demographic and clinical data, including BMI, waist circumference, body fat, blood pressure, fasting plasma glucose, HbA1c, lipid profile, 3-day food diary, International Physical Activity Questionnaire (IPAQ-C), and the sense of fullness will be collected.

On the 12th week, data about the BMI, waist circumference, body fat, blood pressure, fasting plasma glucose, HbA1c, lipid profile, 3-day food diary, IPAQ-C, and the sense of fullness and a questionnaire on the evaluation process will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. BMI >25.0 kg/m2;
2. Waist circumference > 90 cm for men and > 80 cm for women;
3. Aged eighteen years or older;
4. Chinese ethnicity;
5. Can be contacted by telephone;
6. Have the ability to read and understand Chinese; and
7. Can provide informed consent.

Exclusion Criteria:

1. Concurrently participating in any other clinical trials;
2. Concurrently participating in weight control programs;
3. Concomitant intake of weight reduction drugs;
4. Use of calorie restricted diet or specialized diets which contraindicated with low GI diet;
5. Have gastrointestinal problems that would prevent them from following the prescribed diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) | baseline and 12th week
  within- and between-participant changes in BMI, BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m^2, resulting from body mass in kilograms(kg) and body height in metres(m).The body mass and body height will be assessed using an electronic scale and a wall-mounted stadiometer, respectively.

SECONDARY OUTCOMES:
waist circumference | baseline and 12th week
  within- and between-participant changes in waist circumference. Waist circumference will be measured by using the midway point between the top of the hip bone and base of the ribs as a landmark in centimeters(cm) on bare skin at the end of a normal expiration, with arms relaxed at the sides
body fat | baseline and 12th week
  within- and between-participant changes in body fat. Body fat percentage (%) and different body compositions (visceral fat, subcutaneous whole body, subcutaneous trunk, subcutaneous arms, subcutaneous legs) will be assessed by body composition analyser based on the principles of bioelectrical impedance
blood pressure | baseline and 12th week
  within- and between-participant changes in blood pressure. Blood pressure is measured in terms of the systolic pressure over diastolic pressure and is measured in millimeters of mercury (mmHg)
fasting plasma glucose | baseline and 12th week
  within- and between-participant changes in fasting plasma glucose. Fasting plasma glucose will be drawn by venipuncture after an eight-hour overnight. fast for laboratory testing. Fasting plasma glucose is measured in millimoles per liter (mmol/L)
Hemoglobin A1c (HbA1c) | baseline and 12th week
  within- and between-participant changes in HbA1c. HbA1c will be drawn by venipuncture after an eight-hour overnight fast for laboratory testing. HbA1c will be measured in percentage (%)
Total cholesterol (TC) | baseline and 12th week
  within- and between-participant changes in Total cholesterol (TC). It will be drawn by venipuncture after an eight-hour overnight fast. It will be measured in millimoles per liter (mmol/L)
HDL-cholesterol (HDL-C) | baseline and 12th week
  within- and between-participant changes in HDL-cholesterol (HDL-C). It will be drawn by venipuncture after an eight-hour overnight fast. It will be measured in millimoles per liter (mmol/L)
LDL-cholesterol (LDL-C) | baseline and 12th week
  within- and between-participant changes in LDL-cholesterol (LDL-C) level. It will be drawn by venipuncture after an eight-hour overnight fast. It will be measured in millimoles per liter (mmol/L)
Triglycerides level (TG) | baseline and 12th week
  within- and between-participant changes in triglycerides level (TG). It will be drawn by venipuncture after an eight-hour overnight fast. It will be measure in millimoles per liter (mmol/L)
dietary glycemic index (GI) value | baseline and 12th week
  within- and between-participant changes in dietary GI value. The dietary GI value for each participant will be calculated by summing the products of the percentage contribution of each individual food to daily available carbohydrate intake multiplied by the food's GI value.
dietary glycemic load | baseline and 12th week
  within- and between-participant changes in dietary glycemic load. The dietary GL will be calculated by multiplying the dietary GI by the total amount of daily available carbohydrate intake. Dietary will be measured as g per 1000 kcal
calories | baseline and 12th week
  within- and between-participant changes in calories [kcal] intake
carbohydrates | baseline and 12th week
  within- and between-participant changes in carbohydrates[g] intake
fat | baseline and 12th week
  within- and between-participant changes in fat [g] intake
proteins | baseline and 12th week
  within- and between-participant changes in proteins[g] intake
fiber | baseline and 12th week
  within- and between-participant changes in fiber[g] intake
the sense of fullness as dietary satiety | baseline and 12th week
  within- and between-participant changes in the sense of fullness as dietary satiety. The sense of satiety with diet will be assessed by a visual analogue scale (VAS) consisting of a 100mm long line with the left anchor representing "very hungry" and the right anchor representing "very full." The satiety premeal, postmeal and 2 hours postmeal will be measured.

OTHER OUTCOMES:
International Physical Activity Questionnaire (IPAQ-C) | baseline and 12th week
  9 items among four domains on the health-related physical activity. A summary score of metabolic equivalent task/min per week and a categorical score of physical activity (low, moderate and high) will be used to determine the physical activity level of the participants. Physical activity are categories three level: low, moderate and high
self-administer questionnaire | 12th week
  process evaluation with open-ended questions to identify the acceptability, perceived barriers and experience of low GI diet from participants' perspective

CONTACTS AND LOCATIONS:
Overall Officials: Sek Ying Chair, Study Director — The Nethersole School of Nursing, The Chinese University of Hong Kong
Locations (1):
- District Councilor Office, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung LY, Sit JWH, Gao R, Chair SY. Effects of a culturally tailored low-glycaemic index dietary educational intervention on reducing cardiometabolic risk among Chinese adults with obesity: a randomized controlled trial. Eur J Cardiovasc Nurs. 2024 Oct 21;23(7):789-799. doi: 10.1093/eurjcn/zvae062. PMID 38726646